CLINICAL TRIAL: NCT01806532
Title: Regional Lung Inflammation and Expansion in Mechanically Ventilated Patients - a PET/CT Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Marcos Vidal Melo, Associate Professor, Harvard University, Massachusetts General Hospital
Other Study IDs: 2008P000561
Record Dates: First submitted 2013-03-05; First posted 2013-03-07 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Respiratory Failure
Keywords: computed tomography and positron emission tomography; respiration, artificial; respiratory distress syndrome, adult
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Aspiration; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be drawn and plasma stored for future potential biomarker studies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 18F-FDG PET-CT: A total of 10 patients with acute respiratory distress syndrome (ARDS) will be imaged with 2-18F-fluoro-2-deoxy-D-glucose (18F-FDG) and PET-CT scan.

SUMMARY:
The goal of this study is to investigate acute respiratory distress syndrome (ARDS) and septic lung with positron emission tomography (PET) imaging and to examine the distribution of inflammation, as measured by neutrophil metabolic activity.

ELIGIBILITY:
Inclusion Criteria:

Group 1

* Mechanically ventilated patients scheduled to undergo a CT scanning for their routine clinical care
* More than 24 hours of mechanical ventilation
* Less than 15 days of mechanical ventilation if patient presents ALI/ARDS (in order to exclude the late, fibrotic, stage of ARDS)

Group 2

* Mechanically ventilated patients with a diagnosis of sepsis
* Less than 96 hours of mechanical ventilation

Exclusion Criteria:

* Age less than 18 years
* Hemodynamic instability, defined as: systolic blood pressure (SBP) < 90 mmHg that is not adequately stabilized by vasopressors or inotropic agents. For these purposes, SBP will not be considered "adequately stabilized" if the dose of the vasopressor/inotrope has not been stable for at least one hour
* Hypoxemia, defined as: PaO2 < 70 mmHg on an inspired oxygen fraction (FiO2) greater than or equal to 0.9; FiO2 greater than or equal to 0.8 at baseline
* Hemodynamic and/or respiratory instability (as defined, respectively, in 2 and 3), that develop when the patient is mobilized during routine nursing care such as repositioning/washing the patient or changing their bed linens
* Hemodynamic and/or respiratory instability (as defined, respectively, in 2 and 3), that develop when a 15-25 second respiratory pause is introduced as per the study protocol. This will be tested by inducing such a pause prior to transporting the patient
* Patients must be deemed by the treating clinical staff to be able to tolerate leaving the ICU for 90 minutes (40-60 minute imaging time + 30 minute safety margin). Treating MD, RT, and RN must all agree that the patient is stable for transport
* Any acute or chronic condition which, in the opinion of the investigator, might confound the imaging measurements (such as, but not limited to, severe bronchospasm, pulmonary infection, and lung tumor)
* "Air leaks" requiring tube thoracostomy (e.g., pneumothorax, bronchopleural fistula)
* Pregnancy (since this is a study which would expose a fetus to radiation risk)
* Patients who have neither an arterial nor a central venous line at the time of the enrollement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult intensive care patients requiring mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2008-01; Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Regional 18F-FDG activity | Day of imaging.
  Each patient will undergo PET-CT scans and the regional 2-18F-fluoro-2-deoxy-D-glucose (18F-FDG) activity will be measured. This is a measure of regional neutrophil metabolic activity and is used to assess inflammation in the lung. The degree of inflammation will be related to the regional expansion of the lung, as measured by CT scan.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States